CLINICAL TRIAL: NCT03151694
Title: Foundational Work for a Brain-to-Society Diagnostic for Prevention of Childhood Obesity and Its Chronic Diseases Consequences
Brief Title: Brain-to-Society Diagnostic for Prevention of Childhood Obesity and Chronic Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGill University (Other)
Collaborators: The INCLEN Trust International (Unknown)
Responsible Party: Sponsor
Other Study IDs: 227856
Record Dates: First submitted 2017-05-02; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: childhood obesity; body weight; nutritional risk
MeSH Terms: conditions — Obesity; Pediatric Obesity; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA saliva samples were collected for healthy participants between the ages of 6 and 12 years old before proceeding with genotyping of the 7-repeat risk allele on dopamine-4 receptor (DRD4) gene.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DRD4 and DRD2 Polymorphism Detection: The genetic component of endophenotype for responsiveness to environment (ERE) will be characterized with reference to Taq1A allele in dopamine-2 receptor (DRD2) gene and the exon 3 7-repeat allele of the dopamine-4 receptor (DRD4) gene. This will assist in understanding the role of DRD2 and DRD4 in shaping the neurocognitive functions and link to the eating behaviors of the children and other primary outcome variables.

SUMMARY:
This multi-national program applies a breakthrough approach to childhood obesity called, Brain-to-Society (BtS) Diagnostic Approach. In Montreal, Canada and Palwal, India, the investigators will recruit two cohorts of 612 children (6 to 12 years; 306 boy/306 girls) where Whole-of-Society (WoS) transformations are taking place (industrialized societal context with peaking childhood obesity and where a broad governmental plan to promote healthy lifestyle has been adopted -Canada; developing societal context with increasing childhood obesity if replication of past pathways that have lead to double burden; India) are taking place along with World Health Assembly (WHA) resolution A63-12 for marketing of food to children. Individual-level BtS Diagnostic will examine the degree to which individual differences in genetics and biology and differences in the environmental exposures modulate the behavioral, body weight/fatness and nutritional risk over time in the context of WoS transformations. Societal-level BtS Diagnostic shall examine the influence of decisions in policy, investment, business and innovation made by different stakeholders (government, private sector, civil society in health and non-health society systems including agriculture, business and media practices) on the community.

ELIGIBILITY:
Inclusion Criteria:

* Sample population that are exposed to multi-level Whole-of-Society transformation (i.e., Quebec Governmental Action Plan (PAG) and World Health Assembly (WHA) resolution for Quebec sample; Intense Urbanization and Industrialization (IUI) and WHA resolution in India).

Exclusion Criteria:

* first cousin relations were excluded from the sample population.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In two field settings, Canada (Montreal) and India (Palwal), two cohorts of 612 children (6 to 12 years; 306 boy/306 girls) were recruited. Only one child per family was recruited.
Sampling Method: Non-Probability Sample
Enrollment: 1224 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Individual-level BtS Diagnostic 1 | 2 years
  Genotyping and detection of the Taq1A allele in the dopamine-2 receptor (DRD2) gene.
Individual-level BtS Diagnostic 2 | 2 years
  Genotyping and detection of the exon 3 7-repeat allele of the dopamine-4 receptor (DRD4) gene.

SECONDARY OUTCOMES:
Behavioral Assessment | 2 years
  Assess behavior of each participant in relation to food choice
Body Weight Assessment | 2 years
  Assess body weight of each participant
Nutritional Risk Assessment | 2 years
  Assess nutrition intake for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Laurette Dubé, Ph.D., Principal Investigator — McGill University
Locations (2):
- McGill Centre for the Convergence of Health and Economics (MCCHE), Montreal, Quebec, Canada
- The INCLEN Trust International, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Peer-Reviewed Article — http://onlinelibrary.wiley.com/doi/10.1111/jcpp.12646/full
- Available data/document: Peer-Reviewed Article — http://jamanetwork.com/journals/jamapediatrics/fullarticle/2529982
- Available data/document: Peer-Reviewed Article — http://jamanetwork.com/journals/jamapediatrics/fullarticle/2529983